CLINICAL TRIAL: NCT02353585
Title: A Registry of Novel Oral AntiCoagulants and Vitamin K-antagonists In Stroke Patients - a Multi-center Audit Addressing a) Intracerebral Haemorrhage and b) Acute Ischemic Stroke in Patients Treated With Oral Anticoagulants
Brief Title: Novel Oral Anticoagulants in Stroke Patients
Acronym: NOACISP
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ: 2014-027
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Ischemic Stroke; Intracranial Hemorrhages
Keywords: vitamin K-antagonist; novel oral anticoagulants; apixaban; dabigatran; rivaroxaban; edoxaban; direct oral anticoagulants
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intracranial hemorrhage: Intracranial hemorrhage occuring in patients on novel oral anticoagulants (NOAC) or vitamin-K antagonists
- Acute ischemic stroke: Acute ischemic stroke occuring in patients on novel oral anticoagulants (NOAC) or vitamin K antagonists (VKA)

SUMMARY:
The present study will monitor and explore acute neurovascular emergencies in patients treated with NOACs compared to those under treatment with VKAs. The primary aims of this study are: (1) To investigate characteristics, management and outcome of intracranial hemorrhage (ICH) in patients treated with NOAC compared to VKA. (2) To investigate the management and outcome of patients with acute ischaemic stroke under NOAC compared to VKA.

DETAILED DESCRIPTION:
Background: For decades, oral anticoagulation with vitamin K antagonists (VKA) has been the sole option for the treatment of a variety of diseases like venous thrombosis, pulmonary embolism and the prevention of stroke in patients with atrial fibrillation. Despite its clinical efficacy, the treatment with VKA is associated with multiple well-known limitations, including a significant risk of major hemorrhages (especially intracerebral hemorrhage), food and drug interactions, and the need for continued coagulation monitoring for dose control. Recent randomised controlled trials (RCT) have provided promising results with novel oral anticoagulants (NOAC) that do not exhibit the limitations of VKA. Especially for stroke prevention in patients with atrial fibrillation, NOAC have shown comparable or even better protective efficacy while causing less intracerebral hemorrhages (ICH). Eventually, this has led to the marketing approval of Apixaban, Rivaroxaban and Dabigatran for stroke prevention in patients with atrial fibrillation by the Swiss Health Authority (Swissmedic).

Even though the trials reported on the occurrence of acute ischemic strokes or intracerebral hemorrhages in patients under the treatment with NOAC, only limited data and few case reports have been published so far. Thus, aspects concerning the treatment decisions and concepts of management of acute ischemic stroke under NOAC were not addressed in these trials; in particular, the use of acute revascularisation therapies like intravenous thrombolysis (IVT) or intra-arterial treatment (IAT) remains unanswered. Furthermore, characteristics, management and outcome of ICH under the treatment with NOAC were not addressed. Thus, information on relevant aspects of the management of acute neurovascular emergencies under NOACs remains scarce.

Aims: The present study will monitor and explore acute neurovascular emergencies in patients treated with NOACs compared to those under treatment with VKAs. The primary aims of this study are: (1) To investigate characteristics, management and outcome of intracranial hemorrhage (ICH) in patients treated with NOAC compared to VKA. (2) To investigate the management and outcome of patients with acute ischaemic stroke under NOAC compared to VKA.

Methodology: We launch an observational, multi-center (Switzerland and Europe) registry. The leading and coordinating center is located at the Stroke Center of the University Hospital Basel. The following groups of patients admitted to a Stroke Unit of one of the participating centers will be enrolled: A) Patients with ICH occurring while under the treatment with NOAC (last intake <48 hours) or VKA and B) Patients with acute ischaemic stroke occurring while under treatment with NOAC (last intake <48 hours) or VKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ICH occurring while under treatment with NOACs (last intake <48 hours) or VKAs for any indication;
* Patients with acute ischaemic stroke occurring while under treatment with NOACs (last intake <48 hours) or VKAs for any indication.

Exclusion Criteria:

* The patient is, in the opinion of the investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.
* Patients <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the Stroke Unit at the University Hospital Basel (leading and coordinating center).
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Functional neurological outcome | 3 month
  modified Rankin Scale score at 3 month

SECONDARY OUTCOMES:
Hematoma expansion | 0-48 hours
  hematoma expansion on follow-up imaging for patients with intracerebral hemorrhage
symptomatic intracranial hemorrhage | 7 days
  symptomatic intracranial hemorrhage in patients with ischemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Engelter, MD, Principal Investigator — Neurology and Stroke Center; Philippe Lyrer, MD, Principal Investigator — Neurology and Stroke Center
Locations (1):
- Stroke Center, Basel, Switzerland

REFERENCES:
- [Result] Polymeris AA, Meinel TR, Oehler H, Holscher K, Zietz A, Scheitz JF, Nolte CH, Stretz C, Yaghi S, Stoll S, Wang R, Hausler KG, Hellwig S, Klammer MG, Litmeier S, Leon Guerrero CR, Moeini-Naghani I, Michel P, Strambo D, Salerno A, Bianco G, Cereda C, Uphaus T, Groschel K, Katan M, Wegener S, Peters N, Engelter ST, Lyrer PA, Bonati LH, Grunder L, Ringleb PA, Fischer U, Kallmunzer B, Purrucker JC, Seiffge DJ. Aetiology, secondary prevention strategies and outcomes of ischaemic stroke despite oral anticoagulant therapy in patients with atrial fibrillation. J Neurol Neurosurg Psychiatry. 2022 Jun;93(6):588-598. doi: 10.1136/jnnp-2021-328391. Epub 2022 Apr 8. PMID 35396339
- [Derived] Schaub F, Polymeris AA, Schaedelin S, Hert L, Meya L, Thilemann S, Traenka C, Wagner B, Seiffge D, Gensicke H, De Marchis GM, Bonati L, Engelter ST, Peters N, Lyrer P. Differences Between Anticoagulated Patients With Ischemic Stroke Versus Intracerebral Hemorrhage. J Am Heart Assoc. 2022 Jan 4;11(1):e023345. doi: 10.1161/JAHA.121.023345. Epub 2021 Dec 22. PMID 34935409
- [Derived] Seiffge DJ, Kagi G, Michel P, Fischer U, Bejot Y, Wegener S, Zedde M, Turc G, Cordonnier C, Sandor PS, Rodier G, Zini A, Cappellari M, Schadelin S, Polymeris AA, Werring D, Thilemann S, Maestrini I, Berge E, Traenka C, Vehoff J, De Marchis GM, Kapauer M, Peters N, Sirimarco G, Bonati LH, Arnold M, Lyrer PA, De Maistre E, Luft A, Tsakiris DA, Engelter ST; Novel Oral Anticoagulants in Stroke Patients study group. Rivaroxaban plasma levels in acute ischemic stroke and intracerebral hemorrhage. Ann Neurol. 2018 Mar;83(3):451-459. doi: 10.1002/ana.25165. Epub 2018 Mar 3. PMID 29394504
- [Derived] Seiffge DJ, Traenka C, Polymeris AA, Thilemann S, Wagner B, Hert L, Muller MD, Gensicke H, Peters N, Nickel CH, Stippich C, Sutter R, Marsch S, Fisch U, Guzman R, De Marchis GM, Lyrer PA, Bonati LH, Tsakiris DA, Engelter ST. Intravenous Thrombolysis in Patients with Stroke Taking Rivaroxaban Using Drug Specific Plasma Levels: Experience with a Standard Operation Procedure in Clinical Practice. J Stroke. 2017 Sep;19(3):347-355. doi: 10.5853/jos.2017.00395. Epub 2017 Sep 6. PMID 28877563